







Patient Identification Number:

## **CONSENT FORM:**

Title of Project: What difference do chaplains make? An observational study of chaplain interventions in palliative care in UK

Name of Researcher: Professor Austyn Snowden Please initial boxes I confirm that I have read and understood the participant information sheet dated 10-10-2018 for the above study. I have had the opportunity to consider the information provided and had any questions answered satisfactorily. I understand that my participation is voluntary and I can withdraw from the study at any time without giving any notification or reason. I understand that withdrawing from the research study will not incur any adverse consequences to my future treatment. I understand that data already given before my withdrawal will remain in the study. I agree to participate in this research study. I understand that in exceptional circumstances, eg in the event that I disclose potential harm to either myself or others, that my anonymity would be broken and the appropriate authorities contacted. Name of participant Signature of participant Date (Please complete in capital letters) Name of person taking consent Signature of person taking consent Date